CLINICAL TRIAL: NCT01318850
Title: Analysis of the Effects of Cognitive Remediation Therapy on Schizophrenia Patients Through fMRI Techniques
Brief Title: Effects of Cognitive Remediation Therapy on Schizophrenia Patients Through Functional Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: University of Barcelona (Other); Centro de Investigación Biomédica en Red de Salud Mental (Network)
Responsible Party: Principal Investigator, Rafael Penades, Ph.D., Hospital Clinic of Barcelona
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PI070258
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2011-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; cognitive remediation; fMRI
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Training; Coping Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive Remediation Therapy (Experimental): Cognitive Remediation Therapy -Frontal/Executive Program (Delahunty)- (Wykes and Reeder, 2005)
  Interventions: Behavioral: Cognitive Remediation Therapy
- Psychoeducation (Active Comparator): Symptom Management Module from the University of California. Liberman & Kopelowicz (1995)
  Interventions: Behavioral: Psychoeducation
- Healthy Controls (Other): Healthy controls
  Interventions: Other: Healthy controls

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy — The program has a duration of 40 sessions (one hour of duration), with two sessions for week during four months. It is carried out individually and utilizes paper and pencil tasks. The main technique utilized is the scaffolding (to provide strategies when the patient cannot carry out the task and to withdraw him when he is yet able of doing it alone) in a context of learning without errors.
  Other Names: Cognitive training, cognitive enhancement
  Arms: Cognitive Remediation Therapy
Behavioral: Psychoeducation — The program has a duration of 40 sessions (one hour of duration), with two sessions for week during four months. It is carried out individually and utilizes teaching information and coping skills and neuropsychological issues are not addressed.
  Other Names: Coping strategies
  Arms: Psychoeducation
Other: Healthy controls — No intervention
  Other Names: No intervention
  Arms: Healthy Controls

SUMMARY:
Cognitive Remediation Therapy (CRT) can enhance cognitive performance in patients with schizophrenia improving clinical outcome. However, the neurobiological mechanism underlying cognitive improvement is not well understood. The aim of this study is to investigate functional connectivity patterns before and after the neurocognitive rehabilitation therapy, especially in fronto-temporal circuitry.

DETAILED DESCRIPTION:
A controlled randomized study will be carry out with three different groups: patients receiving cognitive rehabilitation treatment (CRT), patients receiving another psychological intervention of control and a healthy control group. A descriptive study of cases will be also carried out. The functional MRI (fRMI) techniques as well as voxel-based morphometry allow individual analysis of cases.

The independent variable is the cognitive rehabilitation treatment. The CRT will be applied according to the manual of Wykes & Reeder (2005) Cognitive Remediation Therapy: Theory and Practice, Ed: Routledge. The program has a duration of 40 sessions (one hour of duration), with two sessions for week during four months. It is carried out individually and utilizes paper and pencil tasks. The main technique utilized is the scaffolding (to provide strategies when the patient cannot carry out the task and to withdraw him when he is yet able of doing it alone) in a context of learning without errors.

The main dependent variable is the functional connectivity cerebral pattern obtained by means of functional magnetic resonance. Other secondary dependent variables are neurocognitive functioning, the symptomatic pattern and the psychosocial functioning obtained from the psychometric evaluation.

All the participants will be evaluated before and after the experimental intervention in neurocognitive areas (Battery will be composed by WAIS-III, RAVLT, Trail Making Test, STROOP color word, WCST, FAS-COWAT), symptomatic area (PANSS) and in social functioning (Social Functioning Scale SFS; Birchwood et al. 1990). The evaluations will be carried out by expert evaluators that will be blind to the experimental distribution. The statistics results analysis will be carry out by means of the statistical package SPSS 15.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to DSM-IV-TR and confirmed by the semi-structured interview (SCID) for the axis 1.
* Presence of cognitive deficit confirmed by the neuropsychological battery.
* Stable symptomatology at least during the last six months and the estimation of not modifying pharmacological antipsychotic treatment.

Exclusion Criteria:

* Presence of organic-cerebral affectation due to neurological or traumatic conditions
* Abuse of psychotropic substances
* Presence of other psychiatric symptomatology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
fMRI patterns of connectivity | Change from baseline in Fractional Anisotropy an Independent Component Analisys indexes at 16 weeks
  Scores on Fractional Anisotropy (FA) index from the Diffusor Technique Images (DTI) and Tract Based Spatial Statistics (TBSS) analyses. Also, scores in the Independent Component Analysis (ICA).

SECONDARY OUTCOMES:
Symptoms | Change from baseline in Positive and Negative Syndrome Scale (PANSS) scores at time 16 weeks
  Scores on Positive and Negative Syndromes Scale (PANSS)
Social Functioning | Change from baseline in scores of Social Functioning Scale at time 16 weeks
  Score on Social Functioning Scale (SFS)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Penadés, Ph.D., Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Penades R, Pujol N, Catalan R, Massana G, Rametti G, Garcia-Rizo C, Bargallo N, Gasto C, Bernardo M, Junque C. Brain effects of cognitive remediation therapy in schizophrenia: a structural and functional neuroimaging study. Biol Psychiatry. 2013 May 15;73(10):1015-23. doi: 10.1016/j.biopsych.2013.01.017. Epub 2013 Feb 26. PMID 23452665
- [Background] Penades R, Pujol N, Catalan R, Masana G, Garcia-Rizo C, Bargallo N, Gonzalez-Rodriguez A, Vidal-Pineiro D, Bernardo M, Junque C. Cortical thickness in regions of frontal and temporal lobes is associated with responsiveness to cognitive remediation therapy in schizophrenia. Schizophr Res. 2016 Mar;171(1-3):110-6. doi: 10.1016/j.schres.2016.01.006. Epub 2016 Jan 15. PMID 26777884